CLINICAL TRIAL: NCT02662439
Title: Role of the Bioimpedance Analysis in Guiding the Diuretic Therapy in Chronic Heart Failure - A Randomized Controlled Trial
Brief Title: Bioimpedance Analysis in Chronic Heart Failure
Status: Suspended | Phase: Not Applicable | Type: Interventional
Sponsor: Peter Studinger (Other)
Responsible Party: Sponsor-Investigator, Peter Studinger, Assistant Professor, Semmelweis University
Organization: Semmelweis University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HF-BCM-15-1
Record Dates: First submitted 2016-01-14; First posted 2016-01-25 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Heart Failure
Keywords: Heart Failure; Bioimpedance analysis; Fluid overload
MeSH Terms: conditions — Heart Failure; Edema

ARMS (2):
- BCM group (Experimental): The patients are measured by Body Composition Monitor (BCM) and both the patient and the physician know the results and adjust the diuretic therapy accordingly.
  Interventions: Device: Body Composition Monitor (BCM)
- Control group (Placebo Comparator): The patients are measured by Body Composition Monitor (BCM) but neither the patient nor the physician know the results, the physician adjusts the diuretic therapy as usual, according to the protocols.
  Interventions: Device: Body Composition Monitor (BCM)

INTERVENTIONS:
Device: Body Composition Monitor (BCM) — In the experimental group, the diuretic therapy adjusted according to the result of the BCM analysis.

SUMMARY:
The aim of this study is to investigate whether the objective measurement of fluid overload by bioimpedance analysis (Body Composition Monitor-BCM) in patient with acute decompensated heart failure would improve the diuretic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with known or newly discovered chronic heart failure admitted to hospital because of the clinical signs of acut cardiac decompensation

Exclusion Criteria:

* High level of fatigue (the patient cannot stand on a scale)
* Amputated upper and/or lower limb(s)
* The BCM analysis is not possible technically (e.g. open wounds on the limbs)
* Severe obesity (>130 kg)
* Patients on chronic hemodialysis or peritoneal dialysis
* Severe fluid volume in the transcellular space
* Patients with a unipolar pacemaker whose sensitivity threshold is very low
* Pregnancy, lactation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Re-hospitalization rate | 12 months

SECONDARY OUTCOMES:
All cause mortality | 12 months

OTHER OUTCOMES:
Quality of life | 3 months
  Measured by validated questionnaire
Renal function decline | 3 months
  Measured by estimated glomerular filtration rate (ml/min/1.73m2)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Studinger, MD, PhD, Principal Investigator — First Department of Medicine, Semmelweis University
Locations (1):
- First Department of Medicine, Semmelweis University, Budapest, Hungary